CLINICAL TRIAL: NCT06277531
Title: Evaluation of diagnostiC Capacity of eccDNAs as Biomarkers in Indetermined biLiary Stricture(ECCBILE): a Prospective Cohort Study
Brief Title: Evaluation of diagnostiC Capacity of eccDNAs as Biomarkers in Indetermined biLiary Stricture(ECCBILE)
Acronym: ECCBILE
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2024086
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Biliary Stricture; Bile Duct Cancer; Pancreas Cancer
Keywords: Malignant Biliary Stricture; Cell-Free Extrachromosomal Circular DNA (eccDNA); Liquid-Biopsies Assay
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — ERCP-obtained bile specimens were centrifuged at 4600 × g for 10 minutes at 4 °C and the supernatants were stored at -80 °C CfDNA was extracted from 0.5 mL of bile specimens and linear DNA was completely digested. For sequencing, after rolling circle amplification, the Nanopore sequencing library for eccDNA was prepared using the ligation sequencing kit and sequenced on a PromethION platform according to the manufacturer's instructions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Biliary stricture is mainly malignant in the adults and caused by several types of fatal malignancies such as pancreatic cancer, cholangiocarcinoma, and metastatic tumor, which have poor prognosis that the overall survival of unresectable lesions is no more than 15 months. The poor outcome often relates to a lack of reliable strategies for early diagnosis, which results in most patients with malignant biliary stricture being already advanced-stage disease at presentation. Therefore, it is critical to discover novel and effective strategies for the early diagnosis of malignant biliary strictures.

Brush cytology and biopsy during endoscopic retrograde cholangiopancreatography (ERCP) are the main methods for recognizing malignant diseases of the bile duct, but their sensitivity is relatively low, 45% and 48.1%, respectively. Even when combined with other biomarkers like carbohydrate antigen 19-9 (CA19-9), their sensitivity is still less than 80%.

In the previous study, the investigators found that bcf-eccDNA has excellent diagnostic value in predicting uncertain bile duct stricture, and the sensitivity and specificity of a related eccDNA in 40 samples are 80.8% and 100%. The sensitivity and specificity of another eccDNA were 92.3% and 92.9%, respectively. However, the sample size is still relatively small, and further prospective studies are needed to evaluate its diagnostic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients is suspected indetermined biliary strictures
* Patients have the indication for ERCP

Exclusion Criteria:

* ERCP failed, or can not obtain bile
* Sever comorbidities
* Predicted overall survival less than 1 year because of other disease
* Patients who are unlikely to comply with the protocol, inability to return for subsequent visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are suspected indetermined biliary strictures
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient is diagnosed with malignant disease from biliary system | in one year
  Malignant tumor is confirmed by histopathology or cytopathology. If the pathology is unclear or inaccessible, 2 gastroenterologists will finally confirm the diagnosis of the bile duct stricture after 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Huang, Principal Investigator — Peking University Third Hospital
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No